CLINICAL TRIAL: NCT02129972
Title: Evaluation of the Video Capsule Colonoscopy for the Detection and the Control of Colon Lesions in Children Presenting Confirmed or Suspected Inflammatory Bowel Disease
Brief Title: Colon Capsule Endoscopy in Children
Acronym: VICCOINBODI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-823
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2018-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease, colon lesions, colon capsule endoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- video capsule endoscopy (Experimental)
  Interventions: Device: Colon videocapsule endoscopy (PillCam colon 2)

INTERVENTIONS:
Device: Colon videocapsule endoscopy (PillCam colon 2) — This is a simple blind (blind for the lecture of the CVC record) study to evaluate the diagnostic value of the colon capsule endoscopy for the detection and the control of colon lesions, the feasibility, tolerance and safety of the CVC compared to the conventional colonoscopy under general sedation in children presented with Inflammatory Bowel Disease.
  Over one week, the patient will undergo two exams (CVC and colonoscopy under general sedation). The exams will be done by two different physicians.
  In order to assess the tolerance, after the completion of both exams, the patients will be asked to answer a "comfort score" questionnaire.
  In order to assess the safety of the CVC, the patients will have a follow-up for adverse events over a 3 weeks period after completion of the CVC and only if the colon video capsule was not recovered during the conventional colonoscopy.
  Other Names: PillCam colon 2

SUMMARY:
The incidence of Inflammatory Bowel Diseases (IBD) is in a continuous progression both in adults as in children. The colonoscopy is considered as the gold standard exam for the diagnosis and the follow-up of the patients presenting or suspected to have an IBD. The follow-up and financial management of this kind of pathology is very much dependent on the quality of the endoscopic images. Because colonoscopy is an expensive and invasive technique which assumes a general sedation, many efforts have been done to develop new less expensive and less invasive techniques in order to offer alternatives to the classic colon endoscopy. One of these new techniques is the colon videocapsule (CVC) endoscopy (PillCam® colon 2 - Given Imaging, Yoqneam, Israel). This is a new promising semi-invasive endoscopic technique which has been successfully validated with adults. We hypothesize that the CVC can be used in children with similar results in terms of efficacy, as is the case for adults.

This prospective simple blind multicenter study, will investigate the diagnostic value of the CVC compared to the conventional colonoscopy under general sedation for the detection and the control of colon lesions in children presenting IBD.

If the feasibility and the efficacy of the colon video capsule technique are also proven for use with children, then this new technique might become a very interesting alternative for the endoscopic examination of the colon because of being less expensive and less invasive.

Moreover, this technique would be very useful as a means of lesions detection all along the digestive tract and not limited to the colon only.

ELIGIBILITY:
Inclusion Criteria:

Will be included in this study are patients:

* Presenting a suspected or confirmed Inflammatory Bowel Disease (IBD) such as Crohn Disease, Ulcerative Colitis or undetermined colitis and who are referred for a conventional colonoscopy;
* Between 8 and 18 years old
* Who are not participating in other clinical trials
* For who a written informed consent was obtained
* Having successfully performed a candy test and the bowel permeability test (using the Patency Alagile ® capsule)

Exclusion Criteria:

Will not be included in this study are patients:

* Presenting a contra indication for colonoscopy under general sedation or for the ingestion of the colon video capsule, especially those for who exist a clinical or radiological suspicion of upper gastrointestinal strictures (esophageal surgery or eosinophil esophagitis) and who presents a dysphagia to solids, swallowing disorders with or without impaired consciousness.
* Who underwent an abdominal surgery during the last 3 months prior to the inclusion visit or who presents signs of bowel stenosis or occlusion
* Who presents a toxic mega colon, radic enteritis, intestinal bowel carcinoma or who receives a chronically non-steroidal anti-inflammatory treatment
* Presenting a contra indication for the bowel preparation agents
* With cardiac pacemaker or other implanted electro medical devices susceptible to interfere with the colon video capsule
* Scheduled for a magnetic resonance imaging (MRI) examination within 7 days following the ingestion of the colon video capsule (and until the evacuation of the capsule has been confirmed) or any other life-threatening conditions

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The diagnostic value of the wireless colon capsule endoscopy | 1 week after the completion of the colon video capsule exam .
  The diagnostic value of the colon video capsule will be estimated based upon the calculated sensitivity of the colon video capsule for the detection and the control of colon lesions in children presented with IBD compared to the colonoscopy sensitivity.

SECONDARY OUTCOMES:
Diagnostic and predictive value of the colon video capsule | 1 week after the completion of the colon video capsule exam
  The diagnostic value expressed by the specificity, positive and negative predictive values of the colon video capsule compared to the results of the colonoscopy under general sedation.
Diagnostic performance of the colon video capsule | 1 week after the completion of both endoscopic exams
  Percentage of the colon lesions successfully detected by the colon video capsule compared to the results recorded during the colonoscopy.
Evaluation of the feasibility and the acceptability by the patient of the colon video capsule compared to the colonoscopy under general sedation | 1 week after the completion of the colon video capsule exam
  Based upon the comfort score calculated after a comfort questionnaire that the patient has been completed after the colon video capsule exam and colonoscopy have been performed
Evaluation of the efficacy of the bowel preparation before the endoscopic examination of the colon | 1 week after the colon video capsule has been performed
  The evaluation will be done using the Boston score.
Descriptive analysis of the visualization and the progression of the colon video capsule over the different segments of the bowel | 1 week after the colon video capsule has been performed
  The analysis will be based upon the description of the different lesions and the time of capsule progression in each bowel segment during the video capsule exam. The different segments will be defined taking into account the anatomic landmarks.

CONTACTS AND LOCATIONS:
Overall Officials: ALAIN LACHAUX, MD, Principal Investigator — HOPITAL FEMME MERE ENFANT CHU DE LYON
Locations (7):
- France (7):
  - Service de Pédiatrie Médicale, Hôpital Pellegrin, CHU de Bordeaux, Bordeaux
  - Service d'Hépatologie, gastroentérologie et nutrition pédiatrique, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Clinique de Pédiatrie, Hôpital Jeanne de Flandre, CHU de Lille, Lille
  - Service de Gastroentérologie, Mucoviscidose et Nutrition, Hôpital Robert Debré, AP-HP, Paris
  - Service de Hépato Gastroentérologie et Nutrition, Hôpital Necker Enfants Malades, AP-HP, Paris
  - Service de Pédiatrie, Hôpital Sud, CHU de Rennes, Rennes
  - Service de Gastroentérologie, Hépatologie, Nutrition et Diabétologie, Hôpital des Enfants, CHU de Toulouse, Toulouse